CLINICAL TRIAL: NCT00376896
Title: A Phase IIa Experimental Medicine Study Assessing Alterations in Regional Cerebral Blood Flow by Functional Magnetic Resonance Imaging (fMRI) in Female IBS Patients and Healthy Controls Following Single Doses of GW876008, a Corticotrophin Releasing Factor 1 Receptor Antagonist (CRF1-RA)
Brief Title: Study On The Effect Of GW876008 On Cerebral Blood Flow In Irritable Bowel Syndrome (IBS) Patients And Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRI103147
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Irritable Colon; Irritable Bowel Syndrome (IBS)
Keywords: IBS fMRI
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — GW 876008

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- GW876008 20mcg (Experimental): GW876008 20mcg
  Interventions: Drug: GW876008 20mcg
- GW876008 200mcg (Experimental): GW876008 200mcg
  Interventions: Drug: GW876008 200mcg
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GW876008 200mcg — GW876008
  Arms: GW876008 200mcg
Drug: GW876008 20mcg — GW876008 20mcg
  Arms: GW876008 20mcg
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
This is a three-period crossover study to compare GW876008 and placebo to see if GW876008 will normalise blood flow responses after different emotional stimuli.

ELIGIBILITY:
Inclusion Criteria:

* The subject should not have been taking and medication for the treatment of IBS for 1 month prior to the study
* Negative serum pregnancy tests (serum a-HCG negative) at Screening (Visit 1), and negative urine pregnancy tests at Visits 1, 2, 3 prior to study medication dose.
* Non-tobacco user (abstinence from tobacco use for at least 1 month before the start of the study).
* Normal electrocardiogram (subjects must have no clinically significant abnormalities on a 12-lead ECG at screen).

Exclusion Criteria:

* Subjects who are pregnant or nursing.
* Current evidence, or history of (at any time in the past) of a biochemical or structural abnormality of the digestive tract. including (but not limited to): inflammatory bowel disease (Crohn's disease or ulcerative colitis); functional dyspepsia; lactose intolerance, not on a stable diet; Celiac Disease
* Subjects who are taking NSAIDs on a regular basis or within 48 hours of a study day.
* The subject has a positive pre-study urine drug/alcohol screen.
* A positive pre-study HIV 1 / 2, Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of the start of the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Signal reductions in the amygdala during viewing of emotional faces and during abdominal pain threat as measured by the fMRI. | throughout the study

SECONDARY OUTCOMES:
Questionnaires to assess IBS symptoms and anxiety | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Dr, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Los Angeles, California, United States